CLINICAL TRIAL: NCT04589494
Title: Comparison Between the Effect of Tramadol Versus Morphine on PD1 and PD1-ligand in Patients With Chronic Cancer Pain
Brief Title: Effect of Tramadol Versus Morphine on PD1 and PD1-ligand in Patients With Chronic Cancer Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Lectruer of anesthesia, ICU and pain manegement, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 493
Record Dates: First submitted 2020-09-14; First posted 2020-10-19 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain
Keywords: morphine; tramadol; PD1 and PD1 ligand
MeSH Terms: conditions — Chronic Pain; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Tramadol; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: tramadol or morphine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tramadol group (Active Comparator): tramadol hydrochloride 100 mg three times daily
  Interventions: Drug: Tramadol Hydrochloride
- morphine group (Active Comparator): morphine 30 mg twise times daily
  Interventions: Drug: Tramadol Hydrochloride

INTERVENTIONS:
Drug: Tramadol Hydrochloride — tramadol hydrochloride 100 mg three times daily , morphine sulphate 30 mg twice daily
  Other Names: morphine sulphate

SUMMARY:
this work is looking for comparison between the effect of tramadol versus morphine on PD1 and PD1-ligand in patients with chronic cancer pain

DETAILED DESCRIPTION:
The use of opioids is the mainstay in the treatment of many types of chronic pain, including cancer and non-cancer-related pain]. Opioids are known to suppress immune function following both acute and chronic administration; however, they appear to be different according to the schedule of administration as well as the state of the organism. Programmed death-1 (PD-1, also known as CD279) belongs to the CD28 receptor superfamily. It is an inhibitory receptor, and its expression is upregulated on activated leukocytes, resulting in an inhibited immune response. PD-1 interacts with two ligands: programmed death ligand-1 (PD-L1, also referred to as B7-H1) and programmed death ligand-2 (PD-L2, also known as B7-DC). PD-L2 is expressed mainly on activated dendritic cells (DCs) and macrophages, whereas PD-L1 is distributed widely. In addition to immune cells, some subsets of tumor cells also express PD-L1 to escape from immunosurveillance. It has been reported that the PD-1/PD-L1 pathway could be activated by surgical stress.

ELIGIBILITY:
Inclusion Criteria:

* patients with cancer pain of varying etiology,
* documented metastatic cancer, currently on step I WHO ladder and whose pain necessitates a shift to step II,
* those who have never received radiotherapy, chemotherapy, or immunosuppressive drugs, -- and in good general and nutritional condition and without infectious diseases at the time of investigation.

Exclusion Criteria:

* abnormal hepatic, renal, and pulmonary function, gastrointestinal pathology, and
* those with cerebral metastases and/or psychological disorders,
* patients with contraindication to morphine or tramadol according to their respective data sheets, and
* patients who could not complete the diary information correctly.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
changes in PD1 and PD1ligand | baseline(0), day15 , day 30
  this is flow cytomertic analyses to the human peripheral blood mononuclear cells (PBMCs) will be separated with a Ficoll-Isopaque density gradient. Flow cytometric analyses will be carried out immediately.

SECONDARY OUTCOMES:
pain assessment | baseline(0), day15 ,day 30
  patient describ his pain severty from 0= no pain to 10= the most sever pain

CONTACTS AND LOCATIONS:
Overall Officials: Shereen M Kamal, Associate Professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt